CLINICAL TRIAL: NCT01563562
Title: A Single-Dose, Open-Label Pharmacokinetic Study of Bardoxolone Methyl in Subjects With Mild, Moderate, and Severe Hepatic Impairment and Normal Hepatic Function
Brief Title: Single-Dose, Open-Label Pharmacokinetic Study of Bardoxolone Methyl in Subjects With Mild, Moderate, and Severe Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1002
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — bardoxolone methyl

ARMS (1):
- Bardoxolone Methyl 20 mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl

INTERVENTIONS:
Drug: Bardoxolone Methyl — Oral, Single dose

SUMMARY:
The purpose of this study is to assess the pharmacokinetic profile of bardoxolone methyl following a single oral dose of 20 mg bardoxolone methyl in subjects with mild, moderate, and severe hepatic impairment, as compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

  1. Male or female subjects between 18 and 70 years, inclusive; must meet all of the following criteria to be included in the study:
  2. Willing to practice method of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested;
  3. Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum pregnancy test result before enrollment into the study;
  4. Body mass index (BMI) between 18 and 37 kg/m2;
  5. Willing and able to give written informed consent for study participation;
  6. Willing and able to cooperate with all aspects of the protocol.

     Subjects with hepatic impairment
  7. Have documented evidence of hepatic cirrhosis by biopsy, nuclear scan, CT, MRI, ultrasound, or other clinically acceptable methods; must meet all of the following criteria to be included in the study:
  8. Be classified as Child-Pugh class A (mild), B (moderate), or C (severe). (See Appendix A for Child-Pugh system.)

Exclusion Criteria:

* All subjects

  1. Participated in another clinical trial of an investigational drug (or a medical device) within 30 days of Study Day -1, or are currently participating in another trial of an investigational drug (or a medical device); with any of the following conditions or characteristics must be excluded from the study:
  2. Known hypersensitivity to any component in the formulation of the study drug, bardoxolone methyl;
  3. Any medical or dental procedure, no matter how minor, that is planned or anticipated to occur during the conduct of the study;
  4. History of drug or alcohol abuse or dependence within the last year;
  5. Donation or receipt of blood or blood components within the 4 weeks prior to Study Day -1. The investigator should instruct subjects who participate in this study not to donate blood or blood components for 4 weeks after the completion of the study;
  6. Abnormal screening ECG which is interpreted by the investigator to be clinically significant;
  7. A positive test for drug(s) of abuse (ethanol, amphetamines, benzodiazepines, barbiturates, cocaine, opiates, or cannabinoids) at the screening or the Day -1 visit, unless the positive drug screen is for a subject with hepatic impairment for a prescription drug and is approved by the principal investigator;
  8. Female subjects who are planning a pregnancy or are pregnant or lactating;
  9. Deemed by the investigator to be inappropriate for this study, including subjects who are unable to communicate with the investigator due to language problems, poor mental development, or impaired cerebral function;
  10. Any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the subject while involved in the study or could potentially influence the study outcome;
  11. Positive test results for human immunodeficiency virus type 1 or 2 antibody at screening;
  12. Have an estimated creatinine clearance < 60 mL/min on Study Day -1 using the Cockcroft-Gault equation (Appendix B);
  13. Any condition possibly affecting absorption, distribution, metabolism or excretion of drugs that may confound the analyses conducted in this study (for example: previous surgery on the gastrointestinal tract that includes removal of parts of stomach, bowel, liver, gall bladder, pancreas, venacaval shunts, or transjugular intrahepatic portosystemic shunts]).

      Subjects with hepatic impairment
  14. Sustained systolic blood pressure > 160 mmHg or < 100 mmHg or a diastolic blood pressure > 100 mmHg at screening or baseline measured after 5 minutes in a sitting position; who have any of the following conditions or characteristics must be excluded from the study:
  15. A pulse rate at rest in a sitting position of < 45 bpm or > 105 bpm;
  16. Documented evidence of primary biliary cirrhosis;
  17. Evidence of recent (two months or less) or current gastrointestinal bleeding;
  18. Platelet counts <50,000 or >450,000.

      Subjects with normal hepatic function
  19. Sustained systolic blood pressure > 150 mmHg or < 100 mmHg or a diastolic blood pressure > 95 mmHg at screening measured after 5 minutes in a sitting position; who have any of the following conditions or characteristics must be excluded from the study:
  20. A pulse rate at rest in a sitting position of < 45 bpm or > 100 bpm;
  21. Evidence or history of or concurrent clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dose administration), hematological, endocrine, immunological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease that in the judgment of the investigator could potentially either pose a health risk to the subject during the study or influence the study outcome;
  22. Evidence of hepatic or biliary dysfunction including elevation of total bilirubin, direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), or alkaline phosphatase levels to greater than the upper limit of normal (ULN);
  23. Positive test results for hepatitis B virus antibody, or hepatitis C virus antibody at screening;
  24. Use of or need for any systemic drug(s) including vitamins or herbal preparations other than drugs used for contraception, within 10 days before Study Day -1 or during the study;
  25. Use of aspirin, non-steroidal anti-inflammatory agents, or acetaminophen within 5 days prior to the ingestion of the study drug; use of aspirin or non-steroidal anti inflammatory agents (but not acetaminophen) will be allowed for isolated episodes of pain at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | 0, 0.5,1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 264, 312, and 360 hours following dose administration

SECONDARY OUTCOMES:
Time to maximum observed concentration | 0, 0.5,1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 264, 312, and 360 hours following dose administration
Oral clearance | 0, 0.5,1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 264, 312, and 360 hours following dose administration
Terminal half-life | 0, 0.5,1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 264, 312, and 360 hours following dose administration
Terminal rate constant | 0, 0.5,1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216, 264, 312, and 360 hours following dose administration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Miami School of Medicine, Miami, Florida
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/